CLINICAL TRIAL: NCT06093633
Title: A Prospective Study to Evaluate the WatchPAT in Comparison to Polysomnography (PSG) Gold Standard in Patients Suspected of Sleep Disorders
Brief Title: A Prospective Study to Evaluate the WP in Comparison to PSG in Patients Suspected of Sleep Disorders
Status: Recruiting | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-001
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Sleep Disorder
Keywords: WatchPAT; Polysomnography; ambulatory device; sleep apnea; apnea-hypopnea index
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The current study is a prospective blinded study to collect data regarding the performance of the WP device in detecting sleep disorders. For that purpose, the WP with finger probe and chest sensor will be worn by the subject simultaneous to PSG in a sleep study at the clinical sleep lab. A PSG system will be recording the PSG data.

DETAILED DESCRIPTION:
Subjects suspected of having sleep disorders who are referred to a sleep study will be screened for potential participation in the study, according to the inclusion and exclusion criteria. Additionally, patients with comorbidities associated with central sleep apnea may be referred from cardiology related divisions, and screened for participation in the study. Recruited patients will be asked to sign an informed consent form. Subject demographic and medical information will be acquired from the subject himself and/or from the subject's medical chart and will be recorded on the appropriate case report forms.

The subjects will be admitted to the clinical sleep laboratory for one night, during which they will undergo conventional full night PSG recording with the standard PSG channels. The WP with finger probe and chest sensor will be worn by the subject simultaneous to PSG. A PSG system will be recording the signals and manual scoring will be performed blinded - without access to WP data. The WP analysis will be done automatically.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-99
* Subjects that are able to read understand and sign the informed consent form of the study or by parents of subjects that are less than 18 years of age that are referred to undergo an overnight sleep study in the clinical sleep laboratory
* Subjects suspected of having sleep disorders or with comorbidities relevant to central sleep apnea.

Exclusion Criteria:

* Permanent pacemaker: atrial pacing or VVI without sinus rhythm.
* Finger deformity that precludes adequate sensor appliance.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with suspected sleep disorders or patients with comorbidities that increase the likelihood of central sleep apnea who are referred for a sleep study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Apnea- Hypopnea Index (AHI) | one night of sleep
  Compares the results of the automatically scored AHI of the WP to the manually scored AHI of the PSG (Gold Standard). AHI is the average number of apnea and hypopnea events per hour of sleep
Sleep Stages | one night of sleep
  Compares the results of the automatically scored sleep stages of the WP to the manually scored sleep stages of the PSG (Gold Standard). Stages are light sleep, deep sleep, REM or Wake.

SECONDARY OUTCOMES:
Respiratory Disturbance Index (RDI) | one night of sleep
  Compares the results of the automatically scored RDI of the WP to the manually scored RDI of the PSG (Gold Standard). RDI is the average number of respiratory events per hour of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Rivi Tauman, Prof,, Principal Investigator — Tel Aviv Medical Center
Locations (3):
- United States (2):
  - Johns Hopkins Bayview Asthma and Allergy Center, Baltimore, Maryland
  - University of Maryland St. Joseph Medical Group, Pulmonary Care & Sleep Medicine, Towson, Maryland
- Tel-Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No